CLINICAL TRIAL: NCT04820179
Title: Phase II Trial Evaluating the Safety and Efficacy of Atezolizumab in Combination With Cabozantinib for the Treatment of Metastatic, Refractory Pancreatic Cancer
Brief Title: Atezolizumab + Cabozantinib in Patients w/ Metastatic, Refractory Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2108097176
Record Dates: First submitted 2021-03-22; First posted 2021-03-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — cabozantinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cabozantinib 40mg + Atezolizumab 1200mg (Experimental): Cabozantinib 40 mg, tablets, oral administration, once daily, continuously. Atezolizumab 1200 mg, administered intravenously, on Day 1 of every 21 day cycle.
  Interventions: Drug: Cabozantinib + Atezolizumab

INTERVENTIONS:
Drug: Cabozantinib + Atezolizumab — All the subjects will be treated with the combination of cabozantinib and atezolizumab until disease progression, unacceptable toxicity or patient consent withdrawal (whichever occurs first).

SUMMARY:
Pancreatic cancer is one of the leading causes of cancer deaths in the United States with limited treatment options, especially for those patients with metastatic disease. Combination treatment with cabozantinib and atezolizumab, has demonstrated safety for the treatment of other cancers and has shown promise in preclinical studies utilizing patient derived pancreas organoids. In this study, patients with refractory, metastatic pancreatic cancer will receive combination cabozantinib + atezolizumab and the efficacy of this treatment will be assessed through overall response rate (ORR), disease control rate (DCR), median overall survival (mOS), and median progression free survival (mPFS). Safety and tolerability of combination cabozantinib plus atezolizumab in metastatic pancreatic cancer patients will also be assessed and immune profiling pre- and post-treatment will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV pancreatic adenocarcinoma, confirmed by histology or cytology. (Note: the primary pancreatic adenosarcoma must be confirmed by histology or cytology. The stage IV metastatic disease does not necessarily need to be confirmed by histology or cytology).
2. Clinical and/or radiographic progression on and/or intolerance to and/or ineligibility for treatment with at least one of the following: a fluoropyrimidine or gemcitabine based chemotherapy treatment regimens
3. Radiographically measurable disease by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Images (MRI or CT Scan) must be completed within 28 days prior to treatment start.
4. Age ≥ 18 years
5. Patients who progress on adjuvant treatment and develop metastatic disease within < 6 months of adjuvant therapy will be considered as having one prior line of treatment and may be eligible pending subject meeting all other inclusion/exclusion criteria.
6. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

   1. Absolute neutrophil count (ANC) ≥ 1500/µL without granulocyte colony-stimulating factor support.
   2. White blood cell count ≥ 2500/µL
   3. Platelets ≥ 100,000/µL without transfusion.
   4. Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
   5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN) with the following exceptions:

      Patients with documented liver metastases: AST and ALT ≤ 5 x ULN Patients with documented liver or bone metastases: ALP ≤ 5 x ULN
   6. Total bilirubin ≤ 1.5 x ULN (for subjects with Gilbert's disease ≤ 3 x ULN).
   7. Serum albumin ≥ 2.8 g/dl
   8. (PT)/INR or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN
   9. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 40 mL/min using the Cockcroft-Gault equation:

      Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72) Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
   10. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h urine protein ≤ 1 g
7. For patients receiving therapeutic anticoagulation, they must have a stable anticoagulant regimen.
8. No clinically significant hypertension as per treating physician or if hypertension, adequate control with anti-hypertensives
9. Negative hepatitis B surface antigen (HBsAg) test at screening
10. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test must be performed for patients who have a positive HCV antibody test.
11. ECOG performance status ≤ 1
12. Recovered to baseline or to CTCAE v5.0 ≤ Grade 1 treatment-related toxicity from prior therapies
13. At least two weeks since last dose of prior treatment
14. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 6 months after the last dose of study treatment.
15. Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating (FSH) level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examinations, or medical history interview by study site.
16. Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

1. Prior treatment with cabozantinib.
2. Prior treatment with atezolizumab and/or CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
3. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 28 days before first dose of study treatment.
4. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 2 weeks before first dose of study treatment.
5. Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
7. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

   1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
   2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
8. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a) Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.

   ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.

   iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.

   iv. Subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #6) for at least 1 week before first dose of study treatment.

   b) Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.

   ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment.

   iii. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
9. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
10. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
11. Lesions invading or encasing any major blood vessels.
12. History of leptomeningeal disease
13. Uncontrolled tumor-related pain

    1. Patients requiring pain medication must be on a stable regimen at study entry.
    2. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
    3. Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
14. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures

    a) Patients with indwelling catheters are allowed.
15. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium >ULN)
16. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix III for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

    1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
    2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    i. Rash must cover < 10% of body surface area ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
17. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

    a) History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
18. Active infection requiring systemic treatment with the following exceptions:

    1. Urinary tract infections
    2. HCV on active treatment
19. Patients with SARS-COV-2 infections with the following exceptions:

    a) Recovery from active symptoms 30 days prior to treatment start.
20. Known history of infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or a known positive test for tuberculosis due to tuberculosis infection.
21. Other clinically significant disorders as deemed by the investigator, that would preclude safe study participation.

    1. Serious non-healing wound/ulcer/bone fracture.
    2. Uncompensated/symptomatic hypothyroidism.
    3. Moderate to severe hepatic impairment.
22. Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 4 weeks before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
23. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment [add reference for Fridericia formula].

    Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
24. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
25. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    1. Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained.
    2. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
26. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
27. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
28. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment of within 6 months after the final dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.
29. Inability to swallow tablets.
30. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
31. Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
32. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
33. Prior allogeneic stem cell or solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate or Stable Disease | Participants will be evaluated for response every 3 cycles (each cycle is 21 days) thereafter until disease progression or death from any cause, whichever occurs first (an average of 6 months)
  To evaluate the efficacy of cabozantinib plus atezolizumab in patients with refractory metastatic pancreatic cancer through overall response rate (ORR) changes or stable disease (SD) after 9 weeks of treatment.

SECONDARY OUTCOMES:
Adverse Event | Participants will be evaluated for response every 3 cycles (each cycle is 21 days) thereafter until disease progression or death from any cause, whichever occurs first (an average of 6 months)
  To evaluate the safety of cabozantinib plus atezolizumab in patients with refractory metastatic pancreatic cancer through the recording of adverse events according to CTCAE version 5.0 and summarized using descriptive statistics.
Toxicities | Participants will be evaluated for response every 3 cycles (each cycle is 21 days) thereafter until disease progression or death from any cause, whichever occurs first (an average of 6 months)
  To evaluate the safety of cabozantinib plus atezolizumab in patients with refractory metastatic pancreatic cancer through the recording of a toxicities according to CTCAE version 5.0 and summarized using descriptive statistics.
Disease Control Rate | Participants will be evaluated for response every 3 cycles (each cycle is 21 days) thereafter until disease progression or death from any cause, whichever occurs first (an average of 6 months)
  To assess the disease control rate (DCR) in patients with refractory metastatic pancreatic cancer treated with combination cabozantinib plus atezolizumab.
Survival | Participants will be evaluated for response every 3 cycles (each cycle is 21 days) thereafter until disease progression or death from any cause, whichever occurs first (an average of 6 months)
  To further define survival outcomes of median overall survival (mOS) and median progression free survival (mPFS) in patients with refractory metastatic pancreatic cancer who receive combination therapy with cabozantinib plus atezolizumab.

OTHER OUTCOMES:
T2 Signal | Participants will be evaluated for response every 3 cycles (each cycle is 21 days) thereafter until disease progression or death from any cause, whichever occurs first (an average of 6 months)
  To quantify T2 signal within the tumor using T2 mapping of tumors pre- and post-treatment with combination cabozantinib plus atezolizumab.
Immune System Effects | Baseline, at 9 weeks, at end of treatment (approx. 6 months), and after disease progression (assessed up to 100 months)
  To explore the immune effects of cabozantinib plus atezolizumab in patients with refractory metastatic pancreatic cancer through Immune profiling of tissue and/or blood collected from study participants
Tumor Response | Participants will be evaluated for response every 3 cycles (each cycle is 21 days) thereafter until disease progression or death from any cause, whichever occurs first (an average of 6 months).
  To evaluate tumor response through comparison of quantified apparent diffusion coefficient (ADC) values of baseline and post-treatment with combination cabozantinib plus atezolizumab tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Rachna Shroff, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No